CLINICAL TRIAL: NCT03101605
Title: Impact of E-learning on the Trainees' Ability to Diagnose and Treat Acute Otitis Media Among Children; A Randomized Educational Trial
Brief Title: E-learning on the Trainees' Ability to Diagnose and Treat Acute Otitis Media Among Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Jocelyn Gravel, MD, MSc, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E-learning for ear exam
Record Dates: First submitted 2017-03-24; First posted 2017-04-05 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Ear Infection
MeSH Terms: conditions — Otitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The physicians evaluating the student performances will be blinded to the randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-learning (Experimental): The intervention for this study will be the completion of an original E-learning module on AOM designed by a team of pediatric residents, pediatricians, a pediatric otolaryngologist, a pediatric emergency physician and a pediatric infectious diseases specialist. The module includes interactive sections on anatomy, epidemiology, pathophysiology, microbiology, diagnostic criteria, treatment options and prognosis. A 5 minute video demonstrating appropriate pediatric ear examination techniques is also included in the module. Throughout the module, many examples of ear pathologies captured on video during a previous study. The E-learning module should take 0.5 hr to complete.
  Interventions: Other: e-learning teaching module
- Standard teaching (Other): The control group will receive a 2h lecture on AOM, which is the "standard" teaching method. Given by a pediatrician or a senior pediatric resident, this lecture, using a PowerPoint© presentation support, encompasses clinical cases, notions of anatomy, epidemiology, pathophysiology, diagnostic criteria, treatment options, and prognosis, describes different ear examination techniques, and shows examples of different pathologies.
  Interventions: Other: Standard teaching method

INTERVENTIONS:
Other: e-learning teaching module — As described
  Arms: e-learning
Other: Standard teaching method — As described
  Arms: Standard teaching

SUMMARY:
An e-learning module to teach how to evaluate ears in children was recently designed. The aim of this study is to measure the impact of this e-learning module on the trainees' ability to appropriately diagnose ear infection in clinical setting.

DETAILED DESCRIPTION:
Background and aims: Acute Otitis Media (AOM) is one of the most common infections of childhood and a leading cause for antibiotics prescription. In a previous study performed at a tertiary care pediatric emergency department, residents were found to have as low as a 52% sensitivity and 74% specificity for the diagnosis of AOM. Seeing this as an opportunity for substantial improvement, an e-learning module on AOM intended for medical students was designed. The primary objective of this study is to measure the impact of this e-learning module on the trainees' ability to appropriately diagnose AOM. The secondary objectives are to assess the preferred learning modality, to evaluate if our e-learning module is associated with improved knowledge on AOM and with better retention at 3 weeks.

Methods: This will be a randomized trial performed at a single tertiary care pediatric emergency department. The participants will be third- and fourth-year medical students doing a general pediatrics rotation. The participants will be randomized to completing the e-learning module at the beginning of their rotation or to receive a 2-hour lecture on the topic of AOM. The primary outcome will be ear examination accuracy measured during their shifts at the emergency department. To measure this, participants will be asked to examine a minimum of five children at risk for AOM, defined as 12-60 months old of age with fever or respiratory symptoms. They will be questioned about the presence or absence of AOM in each examined ear. Attending physicians will control all exams and write down their diagnosis. The primary analysis will be the difference in diagnostic accuracies between the trainees who completed the E-learning module and those who received the lecture. A sample size of 80 medical students each examining a minimum of five children would provide a power of 90% and an alpha-value of 0,05 to demonstrate a difference of 15% in the AOM diagnostic accuracies of medical students who have completed an E-learning module on AOM compared with those receiving a standard lecture on the same topic.

ELIGIBILITY:
Inclusion Criteria:

* Third or fourth-year medical students
* Doing their 6-week rotation in general pediatrics at Sainte-Justine Hospital
* Participation at the introductory meeting on the first day of the rotation

Exclusion Criteria:

* No shifts scheduled at the emergency department during general pediatrics rotation
* Student already recruited in a previous rotation
* Student who evaluated less than 10 ears for the study will not be included in the primary analysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Ear exam accuracy | 1 month
  accuracy of diagnosis of acute otitis media in comparison to the diagnosis made by a staff working at the pediatric emergency

SECONDARY OUTCOMES:
Favorite teaching method | 1 month
  preferred learning modality according to the learners
Immediate theoretical knowledge | 1 hour post training
  Total score in a local knowledge evaluation test composed of the interpretation of 15 ear videos and 5 multiple questions on AOM immediately following training
remote theoretical knowledge | 1 month
  Total score in a local knowledge evaluation test composed of the evaluation of 15 ear videos and 5 multiple questions on AOM immediately following training

CONTACTS AND LOCATIONS:
Locations (1):
- Sainte-Justine Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No